CLINICAL TRIAL: NCT03975660
Title: Evaluation of Objective Pain Measurement Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brendan Carvalho, Chief, Division of Obstetric Anesthesia Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University School of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 51101
Record Dates: First submitted 2019-06-01; First posted 2019-06-05 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Pain; Analgesia; Labor Pain
MeSH Terms: conditions — Pain; Agnosia; Labor Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device Calibration and Validation (Experimental): Patients requesting epidural labor analgesia will have pain levels monitored during labor.
  Interventions: Device: Pain Measurement Device

INTERVENTIONS:
Device: Pain Measurement Device — When participants request labor analgesia, the sensors of the pain measurement device (ROPA System [CereVu Medical, Inc. San Francisco, CA] and Edwards Foresight device) will be applied to the forehead and connected to the device. Data recording is then started.

SUMMARY:
This study will attempt to objectively measure pain with an experimental device. The investigators will apply the device to measure patients "pain" due to uterine contractions during routine clinical care to correlate patients verbal pain ratings and analgesia requirements to that measured by the device. A brain oxygenation device, Edwards Foresight, will be used to concurrently to monitor brain oxygenation and hemodynamics, so the relationship between the CereVu ROPA device objective measure of pain and brain oxygenation/hemodynamic changes and patient-reported pain can be determined.

DETAILED DESCRIPTION:
Despite all the progress in our understanding of the basic mechanisms of pain, the gold standard for measuring pain is still a subjective verbal numeric rating scale rating (0-10) obtained from the individual reporting pain. This method is not objective and cannot be used in all patient populations. This study will attempt to objectively measure pain in laboring mothers with a pain measurement device. The investigators aim to 1) see if the pain measurement device (CereVu ROPA) is capable of reflecting different levels of pain ratings in patients in labor having uterine contractions and then changes in pain after receiving different neuraxial techniques for labor pain and to 2) additionally determine the relationship between the CereVu ROPA device, brain oxygenation/hemodynamic changes and patient-reported pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* ASA 1 or 3 +/-E
* Patient requesting epidural labor analgesia
* Good toco tracing (clearly showing contractions at least every 5 minutes)
* Pain score greater than or equal to 3 out of 10 with contractions

Exclusion Criteria:

* History of chronic pain
* History of chronic opioid use
* BMI > 45
* Allergy to sensor adhesive material, local anesthetic or opioids
* Contraindication to neuraxial block
* Patient on magnesium infusion
* Inability to give informed consent or understand English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, MBBCh, FRCA, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Device Calibration and Validation: When participants request labor analgesia, the sensors of the pain measurement device (ROPA System [CereVu Medical, Inc. San Francisco, CA] and Edwards Foresight device) are applied to the forehead and connected to the device. Data recording is then started.
Period: Overall Study
Arm/Group | Device Calibration and Validation
Started | 130
Completed | 130
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Device Calibration and Validation: When participants request labor analgesia, the sensors of the pain measurement device are applied to the forehead and connected to the device. Data recording is then started.
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (5.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44
  Not Hispanic or Latino | 83
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 45
  Black | 2
  Caucasian | 45
  Latin American | 6
  Native American | 1
  Unknown/Not Reported | 31
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130
Skin Pigmentation Fitzpatrick Scale [Count of Participants; unit: Participants] — Type I: always burns, never tans (palest; freckles) Type II: usually burns, tans minimally (light colored but darker than pale) Type III: sometimes mild burn, tans uniformly (golden honey or olive) Type IV: burns minimally, always tans well (moderate brown) Type V: very rarely burns, tans very easily (dark brown) Type VI: never burns (deeply pigmented dark brown to darkest brown) Population: Participants with skin pigmentation data
  Participants
    Type I: number analyzed (Participants) | 127
    Type I | 20
    Type II: number analyzed (Participants) | 127
    Type II | 47
    Type III: number analyzed (Participants) | 127
    Type III | 26
    Type IV: number analyzed (Participants) | 127
    Type IV | 30
    Type V: number analyzed (Participants) | 127
    Type V | 4
    Type VI: number analyzed (Participants) | 127
    Type VI | 0
Skin Tone [Count of Participants; unit: Participants] — Population: Participants with skin tone data
  Participants
    Fair: number analyzed (Participants) | 129
    Fair | 8
    Light: number analyzed (Participants) | 129
    Light | 21
    Light to Medium: number analyzed (Participants) | 129
    Light to Medium | 37
    Medium: number analyzed (Participants) | 129
    Medium | 15
    Medium to Dark: number analyzed (Participants) | 129
    Medium to Dark | 31
    Dark: number analyzed (Participants) | 129
    Dark | 15
    Very Dark: number analyzed (Participants) | 129
    Very Dark | 2
    Deep: number analyzed (Participants) | 129
    Deep | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Self-report Pain Score
Description: Average patient self-reported pain score on 0 to 10 scale (higher scores correspond to more pain)
Time Frame: During labor up to 2 hours after epidural
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
score on a scale | 4.08 (3.33)

2. Primary Outcome: Correlation of Average Device Pain Score to Average Self-report Pain Score
Description: Pearson correlation
Time Frame: During labor up to 2 hours after epidural
Measure: Number; unit: correlation coefficient
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
correlation coefficient | 0.79

3. Primary Outcome: Correlation Between Pain Score and Brain Oxygenation
Description: Pearson correlation between patient self-reported pain score on 0 to 10 scale (higher scores correspond to more pain) and brain oxygenation (0-100%). This outcome will be assessed in part 2 only.
Time Frame: During labor up to 2 hours after epidural
Measure: Number; unit: correlation coefficient
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
correlation coefficient | 0.05

4. Primary Outcome: Correlation Between Pain Score and Noninvasive Blood Pressure
Description: Pearson correlation between patient self-reported pain score on 0 to 10 scale (higher scores correspond to more pain) and hemodynamic parameter noninvasive blood pressure. This outcome will be assessed in part 2 only.
Time Frame: During labor up to 2 hours after epidural
Measure: Number; unit: correlation coefficient
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
correlation coefficient
  Pain score and diastolic blood pressure | 0.20
  Pain score and systolic blood pressure | 0.22

5. Primary Outcome: Correlation Between Pain Score and Heart Rate
Description: Pearson correlation between patient self-reported pain score on 0 to 10 scale (higher scores correspond to more pain) and hemodynamic parameter heart rate. This outcome will be assessed in part 2 only.
Time Frame: During labor up to 2 hours after epidural
Measure: Number; unit: correlation coefficient
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
correlation coefficient | 0.20

6. Primary Outcome: Correlation Between Pain Score and Pulse Oximetry
Description: Correlation between patient self-reported pain score on 0 to 10 scale (higher scores correspond to more pain) and hemodynamic parameter pulse oximetry (Sp02). This outcome will be assessed in part 2 only.
Time Frame: During labor up to 2 hours after epidural
Measure: Number; unit: correlation coefficient
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
correlation coefficient | 0.05

7. Secondary Outcome: Time to Reach Pain Score 2 or Less Out of 10
Description: Pain score on 0 to 10 scale (higher scores correspond to more pain)
Time Frame: within 45 minutes after the block placement
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
minutes | 17.2 (12.60)

8. Secondary Outcome: Time Taken for Pain Device Score to be Below Validated Value
Description: Validated value is from the validated reading recorded by the sensor in the pilot study
Time Frame: within 45 minutes after the block placement
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
minutes | 16.6 (12.22)

9. Secondary Outcome: Patient Reported Pain Scores After Block
Description: Pain score on 0 to 10 scale (higher scores correspond to more pain). Pain scores were obtained at random intervals and the scores were summed and averaged to create the reported score. Patients stopped rating pain once the level dropped to zero.
Time Frame: Up to approximately 45 minutes after the block placement
Population: Participants with data for the respective time frame
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 125
score on a scale
  Participants with data obtained for ≥ 15 minutes | 2.0 (2.50)
  Participants with data obtained for ≥ 30 minutes: number analyzed (Participants) | 92
  Participants with data obtained for ≥ 30 minutes | 2.0 (2.20)
  Participants with data obtained for ≥ 45 minutes: number analyzed (Participants) | 39
  Participants with data obtained for ≥ 45 minutes | 1.0 (1.40)

10. Secondary Outcome: Device Recorded Pain Scores After Block
Description: Device pain score validated measure (range: 0 to 10, higher scores correspond to more pain). Pain scores were obtained at random intervals and the scores were summed and averaged to create the reported score. Device recording was discontinued when pain level dropped to zero.
Time Frame: Up to approximately 45 minutes after the block placement
Population: Participants with data recorded within the respective time frame
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 125
score on a scale
  Participants with data recording ≥ 15 minutes | 2.9 (1.90)
  Participants with data recording ≥ 30 minutes: number analyzed (Participants) | 92
  Participants with data recording ≥ 30 minutes | 2.7 (1.99)
  Participants with data recording ≥ 45 minutes: number analyzed (Participants) | 39
  Participants with data recording ≥ 45 minutes | 1.5 (1.44)

11. Secondary Outcome: Dermatomal Level at 45 Minutes After Block Placement as a Measure of Sensory Blockade Level
Time Frame: 45 minutes
Population: Dermatomal testing was not performed to reduce burden on participants. The study team decided it was not critical prior to the start of the study, however, the study protocol was not amended to reflect this change. No data were collected for this Outcome Measure.
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 0

12. Secondary Outcome: Count of Participants With Block Failures
Time Frame: within 45 minutes after the block placement
Measure: Count of Participants; unit: Participants
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
Participants | 18

13. Secondary Outcome: Count of Participants With Maternal Side Effects
Description: Monitored maternal side effects will include nausea, pruritis, hypotension
Time Frame: within 45 minutes after the block placement
Measure: Count of Participants; unit: Participants
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
Participants | 0

14. Secondary Outcome: Count of Participants With Fetal Side Effects
Description: Monitored fetal side effects include fetal decelerations early/variable/late
Time Frame: within 45 minutes after the block placement
Measure: Count of Participants; unit: Participants
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
Participants | 0

15. Secondary Outcome: Count of Participants Needing Physician Intervention
Time Frame: within 45 minutes after the block placement
Measure: Count of Participants; unit: Participants
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
Participants | 0

16. Secondary Outcome: Time From Epidural to Delivery
Time Frame: from epidural to delivery (average approximately 9 hours)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
minutes | 560 (398)

17. Secondary Outcome: Count of Participants With Normal Vaginal Delivery
Time Frame: from epidural to delivery (expected average: 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
Participants | 109

18. Secondary Outcome: Count of Participants With Assisted Vaginal Delivery
Time Frame: from epidural to delivery (expected average: 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
Participants | 2

19. Secondary Outcome: Count of Participants With Cesarean Delivery
Time Frame: from epidural to delivery (expected average: 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Device Calibration and Validation
Number analyzed (Participants) | 130
Participants | 19

ADVERSE EVENTS:
Time Frame: 1 day (average approximately 2 hours)
Arm/Group | Device Calibration and Validation
All-Cause Mortality (participants affected / at risk) | 0/130
Serious Adverse Events (participants affected / at risk) | 0/130
Other Adverse Events (participants affected / at risk) | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03975660/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT03975660/SAP_001.pdf